CLINICAL TRIAL: NCT02616601
Title: A Multicenter, Randomized, Double-Blind, Vehicle-Controlled, Parallel Group Comparison Study to Determine the Therapeutic Equivalence of Generic Fluorouracil Cream, 0.5% and Carac® (Fluorouracil) Cream, 0.5% in Subjects With Actinic Keratoses
Brief Title: Multicenter, Double-blind, Placebo Controlled Comparing Test Fluorouracil Cream to Carac Cream in Actinic Keratosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Actavis Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 094-8251-301
Record Dates: First submitted 2015-11-25; First posted 2015-11-30 (Estimated); Results first posted 2019-07-17 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-06

CONDITIONS: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic | interventions — Fluorouracil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Generic Fluorouracil Cream (Experimental): Participants are to apply up to 1 gram of generic fluorouracil 0.5% topical cream once daily for 2 weeks as a thin film to the skin of the treatment area and rub until the cream is no longer visible. Participants will be instructed to apply the study drug 10 minutes after thoroughly washing, rinsing, and drying the entire treatment area and 1 to 2 hours before bedtime. Study drug should be left on the skin for approximately 8 hours and then removed by washing the area with mild soap and water. Treatment should be continued for the full treatment course even if the actinic keratoses lesions appear to be gone.
  Interventions: Drug: Generic Fluorouracil Cream
- Carac® (Fluorouracil) Cream (Active Comparator): Participants are to apply up to 1 gram of Carac (fluorouracil) 0.5% topical cream once daily for 2 weeks as a thin film to the skin of the treatment area and rub until the cream is no longer visible. Participants will be instructed to apply the study drug 10 minutes after thoroughly washing, rinsing, and drying the entire treatment area and 1 to 2 hours before bedtime. Study drug should be left on the skin for approximately 8 hours and then removed by washing the area with mild soap and water. Treatment should be continued for the full treatment course even if the actinic keratoses lesions appear to be gone.
  Interventions: Drug: Carac® (Fluorouracil) Cream
- Vehicle Cream (Placebo Comparator): Participants are to apply up to 1 gram of vehicle topical cream once daily for 2 weeks as a thin film to the skin of the treatment area and rub until the cream is no longer visible. Participants will be instructed to apply the study drug 10 minutes after thoroughly washing, rinsing, and drying the entire treatment area and 1 to 2 hours before bedtime. Study drug should be left on the skin for approximately 8 hours and then removed by washing the area with mild soap and water. Treatment should be continued for the full treatment course even if the actinic keratoses lesions appear to be gone.
  Interventions: Drug: Vehicle Cream

INTERVENTIONS:
Drug: Generic Fluorouracil Cream — Topical cream, generic formulation of the brand product.
  Other Names: 5-FU
  Arms: Generic Fluorouracil Cream
Drug: Carac® (Fluorouracil) Cream — Topical cream, brand product.
  Other Names: 5-FU
  Arms: Carac® (Fluorouracil) Cream
Drug: Vehicle Cream — Topical cream, placebo. Has no active ingredient.
  Arms: Vehicle Cream

SUMMARY:
This study is to evaluate the efficacy and safety of a generic formulation of fluorouracil 0.5% cream against the brand product (Carac) in participants with actinic keratoses.

DETAILED DESCRIPTION:
This is a multicenter, double-blind, vehicle-controlled, parallel group comparison study of a generic fluorouracil cream, 0.5% and Carac (fluorouracil) Cream, 0.5% in participants with actinic keratoses on the full face or balding scalp.

ELIGIBILITY:
Inclusion Criteria:

* Participant is male and/or female, 18 years of age or older.
* Participant is willing and able to give written informed consent.
* Participant is willing and able to apply the test article(s) as directed, comply with study instructions and commit to all follow-up visits for the duration of the study.
* Participant has a clinical diagnosis of actinic keratoses with at least 5 and no more than 10 clinically typical, visible or palpable, discrete, actinic keratoses (AK) lesions, each at least 4 millimeters (mm) in diameter on the face (excluding ears) or balding scalp.
* Participant is in good general health and free of any disease state or physical condition that might impair evaluation of AK lesions or which, in the investigator's opinion, exposes the participant to an unacceptable risk by study participation.
* Females must be post-menopausal, surgically sterile, or use an effective method of birth control with a negative urine pregnancy test (UPT) at the Baseline Visit.

Exclusion Criteria:

* Participant is pregnant, lactating, or is planning to become pregnant during the study.
* Participant is currently enrolled in an investigational drug or device study.
* Participant has used an investigational drug or investigational device treatment within 30 days prior to the Baseline Visit.
* Participant has hyperkeratotic, hypertrophic, or large mat-like AK lesions (for example, an AK lesion >1 cm^2 in size) within the treatment area.
* Participant has the need or plans to be exposed to artificial tanning devices or excessive sunlight during the study.
* Participant is immunosuppressed (for example, human immunodeficiency virus (HIV), systemic malignancy, graft host disease)
* Participant has experienced an unsuccessful outcome from previous topical fluorouracil therapy (an unsuccessful outcome is defined as after a reasonable therapeutic study with no compliance issues and the topical drug did not work).
* Participant has a history of sensitivity to any of the ingredients in the test articles.
* Participant has known dihydropyrimidine dehydrogenase (DPD) enzyme deficiency.
* Participant used topical creams, lotions, or gels of any kind within the selected treatment area within 1 day prior to entry into the study.
* Participant has used topical medications; corticosteroids, alpha hydroxy acids (for example, glycolic acid, lactic acid, etc. >5%), beta hydroxy acid (salicylic acid >2%), urea >5%, 5-fluorouracil, diclofenac, imiquimod, ingenol mebutate; or prescription retinoids (for example, tazarotene, adapalene, tretinoin) within the selected treatment area (face or balding scalp) within 1 month prior to the Baseline Visit.
* Participant has had cryodestruction, curettage, photodynamic therapy, surgical excision, or other treatments for AK within the selected treatment area (face or balding scalp) within 1 month prior to the Baseline Visit.
* Participant has used oral corticosteroid therapy, interferon, cytotoxic drugs, immunomodulators, immunosuppressive therapies, or retinoids within 1 month prior to the Baseline Visit.
* Participant has had dermatologic procedures or surgeries such as: laser resurfacing, Psoralen + ultraviolet A (PUVA) therapy, ultraviolet B therapy, chemical peels, or dermabrasion within the selected treatment area (face or balding scalp) within 6 months prior to the Baseline Visit.
* Participant has lesions suspicious for skin cancer (skin cancer not ruled out by biopsy) or untreated skin cancers within the selected treatment area (face or balding scalp).
* Participant has any skin pathology or condition on the face or balding scalp that, in the Investigator's opinion, could interfere with the evaluation of the test article or requires the use of interfering topical, systemic, or surgical therapy.
* Participant has any condition which, in the Investigator's opinion, would make it unsafe or preclude the participant's ability to fully participate in this research study.
* Participant is unable to communicate or cooperate with the Investigator due to language problems, poor mental development, impaired cerebral function, or physical limitations.
* Participant is known to be noncompliant or is unlikely to comply with the requirements of the study protocol (for example, due to alcoholism, drug dependency, mental incapacity) in the opinion of the Investigator.
* Participant has been previously enrolled in the same study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 422 (Actual)
Dates: Start 2015-02-27 (Actual); Primary Completion 2015-09-17 (Actual); Study Completion 2015-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Actavis Inc.
Locations (17):
- United States (17):
  - Investigative Site 2, Fremont, California
  - Investigative Site 16, Los Angeles, California
  - Investigative Site 17, San Diego, California
  - Investigative Site 4, Denver, Colorado
  - Investigative Site 10, Newnan, Georgia
  - Investigative Site 5, Boise, Idaho
  - Investigative Site 1, Arlington Heights, Illinois
  - Investigative Site 11, Buffalo Grove, Illinois
  - Investigative Site 3, Carmel, Indiana
  - Investigative Site 9, Plainfield, Indiana
  - Investigative Site 6, South Bend, Indiana
  - Investigative Site 8, Clinton Township, Michigan
  - Investigative Site 13, Warren, Michigan
  - Investigative Site 12, Fridley, Minnesota
  - Investigative Site 15, Albuquerque, New Mexico
  - Investigative Site 7, High Point, North Carolina
  - Investigative Site 14, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The populations for this study included the Safety Population, the Per-Protocol (PP) Population, and the modified Intent-to-Treat (mITT) population.
Groups:
- Generic Fluorouracil Cream: Participants applied up to 1 gram of generic fluorouracil 0.5% topical cream once daily for 2 weeks (wks) as a thin film to the skin of the treatment area and rub until the cream was no longer visible. Participants were instructed to apply the study drug 10 minutes after thoroughly washing, rinsing, and drying the entire treatment area and 1 to 2 hours before bedtime. Study drug was to have been left on the skin for approximately 8 hours and then removed by washing the area with mild soap and water. Treatment should have continued for the full treatment course even if the actinic keratoses lesions appeared to be gone.
- Carac (Fluorouracil) Cream: Participants applied up to 1 gram of Carac (fluorouracil) 0.5% topical cream once daily for 2 weeks as a thin film to the skin of the treatment area and rub until the cream was no longer visible. Participants were instructed to apply the study drug 10 minutes after thoroughly washing, rinsing, and drying the entire treatment area and 1 to 2 hours before bedtime. Study drug was to have been left on the skin for approximately 8 hours and then removed by washing the area with mild soap and water. Treatment should have continued for the full treatment course even if the actinic keratoses lesions appeared to be gone.
- Vehicle Cream: Participants applied up to 1 gram of vehicle topical cream once daily for 2 weeks as a thin film to the skin of the treatment area and rub until the cream was no longer visible. Participants were instructed to apply the study drug 10 minutes after thoroughly washing, rinsing, and drying the entire treatment area and 1 to 2 hours before bedtime. Study drug was to have been left on the skin for approximately 8 hours and then removed by washing the area with mild soap and water. Treatment should have continued for the full treatment course even if the actinic keratoses lesions appeared to be gone.
Period: Overall Study
Arm/Group | Generic Fluorouracil Cream | Carac (Fluorouracil) Cream | Vehicle Cream
Started | 140 | 140 | 142
Safety Population (Randomized participants who received the study drug.) | 140 | 140 | 142
mITT Population (Randomized participants, applied ≥1 dose study drug, returned for ≥1 post-baseline evaluation visit) | 137 | 136 | 138
PP Population (mITT, >75-125% doses and >6 consecutive doses or discontinued for lack of treatment- completed ≥8wks) | 112 | 121 | 123
Completed | 131 | 136 | 135
Not Completed | 9 | 4 | 7
Not completed — Withdrawal by Subject | 4 | 4 | 3
Not completed — Adverse Event | 2 | 0 | 2
Not completed — Death | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — Non-Compliance with Test Article | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants who received the study drug (Safety Population).
Groups:
- Generic Fluorouracil Cream: Participants applied up to 1 gram of generic fluorouracil 0.5% topical cream once daily for 2 weeks as a thin film to the skin of the treatment area and rub until the cream was no longer visible. Participants were instructed to apply the study drug 10 minutes after thoroughly washing, rinsing, and drying the entire treatment area and 1 to 2 hours before bedtime. Study drug was to have been left on the skin for approximately 8 hours and then removed by washing the area with mild soap and water. Treatment should have continued for the full treatment course even if the actinic keratoses lesions appeared to be gone.
- Total: Total of all reporting groups
Arm/Group | Generic Fluorouracil Cream | Carac (Fluorouracil) Cream | Vehicle Cream | Total
Number analyzed (Participants) | 140 | 140 | 142 | 422
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.7 (9.46) | 67.4 (9.43) | 67.1 (11.13) | 67.4 (10.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 18 | 20 | 54
  Male | 124 | 122 | 122 | 368
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 1 | 4
  Not Hispanic or Latino | 139 | 138 | 141 | 418
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 138 | 140 | 141 | 419
  More than one race | 1 | 0 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment Success (Complete Clearance) at Week 6
Description: Percentage of participants with treatment success (complete clearance) at Week 6 (4 weeks after completion of 2 weeks of treatment). Complete clearance was defined as having no (zero) clinically visible actinic keratoses (AK) lesions in the treatment area at the Week 6/End Of Study visit. All AK lesions (baseline and new lesions) independent of size within the treatment area were treated and included in the efficacy lesion count.
Time Frame: Week 6
Population: Participants in mlTT population who met inclusion/exclusion criteria, applied 75%-125% applications of study drug, did not miss applications for more than 3 consecutive days, no evidence of dosing noncompliance, and completed evaluation at Week 6 within ±4 days with no protocol violations that would affect treatment evaluation (PP Population).
Measure: Number; unit: percentage of participants
Arm/Group | Generic Fluorouracil Cream | Carac (Fluorouracil) Cream | Vehicle Cream
Number analyzed (Participants) | 112 | 121 | 123
percentage of participants | 33.9 | 33.9 | 3.3
Statistical Analysis 1: Comparison: Generic Fluorouracil Cream vs Carac (Fluorouracil) Cream; Test type: Equivalence — If the 90% confidence interval on the percentage difference between generic fluorouracil cream and Carac (fluorouracil) cream lesion clearance were contained within the interval -0.20 to +0.20, and each of these percentages was greater than and statistically different (p<0.05) from the vehicle cream percentage, then generic fluorouracil cream and Carac (fluorouracil) cream were considered to be therapeutically equivalent; Mean Difference (Net) = 0.04, 90% CI 2-sided [-11.03 to 11.11] — 90% Wald's confidence interval with a continuity correction for the difference (Generic Fluorouracil Cream - Carac [Fluorouracil] Cream) in complete clearance rates
Statistical Analysis 2: Comparison: Generic Fluorouracil Cream vs Vehicle Cream; Test type: Superiority; p < 0.0001, Fisher Exact
Statistical Analysis 3: Comparison: Carac (Fluorouracil) Cream vs Vehicle Cream; Test type: Superiority; p < 0.0001, Fisher Exact

ADVERSE EVENTS:
Time Frame: Baseline up to Week 6
Description: Adverse events were collected from participants who were randomized and received the study drug.
Arm/Group | Generic Fluorouracil Cream | Carac (Fluorouracil) Cream | Vehicle Cream
All-Cause Mortality (participants affected / at risk) | 1/140 | 0/140 | 0/142
Serious Adverse Events (participants affected / at risk) | 4/140 | 1/140 | 2/142
Other Adverse Events (participants affected / at risk) | 21/140 | 13/140 | 9/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Generic Fluorouracil Cream (N=140) | Carac (Fluorouracil) Cream (N=140) | Vehicle Cream (N=142)
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Aortic aneurysm (Vascular disorders) | 1 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Inguinal hernia strangulated (Gastrointestinal disorders) | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 0
Aortic stenosis (Vascular disorders) | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Generic Fluorouracil Cream (N=140) | Carac (Fluorouracil) Cream (N=140) | Vehicle Cream (N=142)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1
Eye Irritation (Eye disorders) | 2 (4) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1
Application site dermatitis (General disorders) | 1 | 0 | 0
Seasonal Allergy (Immune system disorders) | 1 | 0 | 0
Cytstitis (Infections and infestations) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0
Acute Kidney Injury (Renal and urinary disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1
Application site erythema (General disorders) | 1 | 0 | 0
Application site pain (General disorders) | 2 | 0 | 0
Application site pruritus (General disorders) | 1 | 0 | 0
Chills (General disorders) | 0 | 0 | 1
Influenza like illness (General disorders) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 3 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 1 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 2 | 2 | 2
Haematuria (Renal and urinary disorders) | 0 | 1 | 0
Hypertonic bladder (Renal and urinary disorders) | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.